CLINICAL TRIAL: NCT02427438
Title: Home Program Education for Patients With Low Back Pain: Does it Matter? A Prospective Study
Brief Title: Home Program Education for Patients With Low Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not recruiting subjects currently
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0672
Record Dates: First submitted 2015-04-22; First posted 2015-04-28 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Low Back Pain; Lumbago; Spinal Instability
Keywords: video; handout; home program; stabilization; strengthening; core
MeSH Terms: conditions — Low Back Pain | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Home Program Education (Active Comparator): Subjects in this group will complete the same 8 weeks of home program exercises for lumbar instability. The home program exercises will be completed using a video with verbal instruction for guidance of proper technique and repetitions.
  Interventions: Other: Video
- Handout Home Program Education (Active Comparator): Subjects will complete the same 8 weeks of home program exercises for lumbar instability. The home program exercises will be completed using a handout with two dimensional pictures and written instructions for guidance of proper technique and repetitions.
  Interventions: Other: Handout

INTERVENTIONS:
Other: Video — A video with moving demonstration and verbal instruction of the exercise to strengthen low back
  Arms: Video Home Program Education
Other: Handout — A handout with a two dimensional picture and written instruction of the exercise to strengthen low back
  Arms: Handout Home Program Education

SUMMARY:
The primary purpose of this study is to assess the effect size of the change in Oswestry Disability Questionnaire (ODQ) score over the 8 week follow-up period between the video based instruction or standard of care hand-out with pictures and written instructions for subjects meeting the clinical prediction rule for lumbar stabilization.

The second purpose will be to determine if there is a subset of physical examination and self-reported variables that are associated with having a successful result (ODQ improvement by at least 6 points) and if the subset of variables are affected by whether or not the subject was in the intervention (video) or control (handout) group.

DETAILED DESCRIPTION:
Approximately fifty percent of patients seeking help in outpatient orthopedic clinics and roughly thirty percent of people will experience some low back pain (LBP) at some time in their life.(1) LBP is the second leading cause of missed days of work per year and results in around ninety billion dollars per year in medical costs. (1) Physical therapy interventions for LBP could include manual therapy, exercise, traction, range of motion, modalities, postural education, or a combination of these interventions.(2-5) Medical treatment for LBP could include medications, imaging, laboratory studies, injections, surgery, or counseling through pain psychology.(6-7) Many research studies are inconclusive regarding effective treatment.

In 1995 a treatment based classification system for patients with acute low back pain was published.(8) Patients were categorized into one of four categories: manipulation, directional exercises (flexion, extension, lateral shift correction), immobilization, or traction. (8)This classification system led to further validation of the categories and clinical prediction rules (CPR) related to best treatment outcomes.(9-11) In 2005, Hicks built upon the initial classification system for immobilization when he published a preliminary CPR identifying which patients were most likely to benefit from lumbar stabilization.(10) Hicks identified the following predictors for patient response to stabilization exercises: individuals younger than age forty, straight leg raise greater than ninety-one degrees, and aberrant motions or a positive prone instability test.(10) Hicks reported a presence of three or more of these variables had a positive likelihood ratio of 4.0 for a 95% confidence interval.(10) However, no studies to date have confirmed such results nor validated this clinical prediction rule.

Home program prescription background Evidence for using video for home program prescription is limited. However, video based home programs have been successfully used for patients with Huntington's disease, traumatic brain injury (TBI), spinal cord injury, brachial plexus injuries, and general shoulder strengthening.(12-15) Medical studies demonstrate that patients comprehend information better when communicated via educational videos as opposed to educational pamphlets about various disorders.(16-18)

Problem Statement:

Currently, there is no literature evaluating the use of video home programs for patients with LBP or identifying who may benefit from this form of clinical education. Home program handouts frequently depict photographs or figures with incorrect form or instructions. Video based home programs demonstrating the stabilization techniques for patients may provide correct form and accurate instructions. With such programs, patient comprehension and technical reproduction of the exercises may improve. Video-based home programs could lead to fewer clinic visits and decreased cost per episode of care.

Given the numerous factors that contribute to limited clinic visits in LBP patients, more effective communication should be beneficial during treatment. We do not know if patient learning styles may influence compliance with varying modes of home exercise program prescriptions. Video based home exercise programs may also be a better fit for patients who are more auditory or visual learners as defined by the Visual, Auditory, Reading, Kinesthetic (VARK) learning inventory. (19) Auditory learners prefer information being transferred by listening. Visual learners prefer maps, charts, and perhaps videos over written charts or instructions.

ELIGIBILITY:
Inclusion Criteria:

1. presence of aberrant movement (Gower's sign, painful arc of motion, poor reversal of lumbopelvic rhythm)
2. Positive prone instability test
3. Straight leg raise greater than ninety-one degrees
4. Age under 40

Exclusion Criteria:

1. Anyone not meeting the 3/4 clinical prediction rules
2. Those unable to access video based exercise instructions
3. A prior spinal fusion, tumor, infection
4. Two or more neurological symptoms such as upper motor neuron signs, myotomal weakness, dermatomal sensory changes, or abnormal reflexes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Questionnaire (ODQ) | 8 weeks
  The ODQ measures level of disability with patients presenting with low back pain. It is also reliable and has excellent construct validity.(10, 34-36) The ODQ will be assessed at baseline and after eight weeks of therapy to determine the overall success of stabilization based treatment on patient function.(10) The Oswestry has ten sections, one to assess pain and the remaining which assesses functional activities. Each section is scored from 0 to 5 which indicates the level of limitation with that given activity. Each score is then totaled and then doubled to give a percentage of disability. Higher scores on the Oswestry indicate greater levels of disability. A five to six point improvement on the Oswestry is considered the minimum clinically important difference with a fifty percent improvement being defined as "success" by Hicks.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 8 weeks
  All subjects will complete a numeric pain rating using the traditional eleven point VAS scale. This will be assessed at every clinic visit. The VAS consists of a 100 mm line in which patients mark their pain on a scale from No Pain to Worst Pain Imaginable. This has been shown to be reliable and valid in prior research studies for low back pain. The VAS also is sensitive in detecting small amounts of change. 24 Prior research demonstrates that the repeatability of the VAS is good with correlation coefficients ranging from 0.97 to 0.99.(25) According to Jenson, the VAS also has greater levels of discrimination when using a 101 point scale.(26) Majority of research articles using the VAS define a statistically significant reduction as 50%.(26)

OTHER OUTCOMES:
Fear and Avoidant Behaviors Questionnaire | 8 weeks
  The Fear and Avoidant Behaviors Questionnaire (FABQ) will be used to screen for psychosocial contributions to a participants pain and function. The FABQ will be assessed at baseline and 8 weeks/discharge. Two subscales within this questionnaire assess physical activity and work. Responses are marked on a 7-point Likert scale ranging from completely disagree to completely agree. Higher scores indicate higher levels or fear-avoidance beliefs on both subscales. The FABQ is reliable and valid for use with LBP patients.27-29 Test retest reliability of the physical activity subscale has been shown to be acceptable at ICC=0.72 to 0.90. (30, 31) Fritz demonstrated that the FABQ work subscale can be used to identify which patients are at risk of not returning to work after four weeks of work-related injury. (32) A clinically important change level has not yet been determined for use of the FABQ. Woby however, demonstrated that changes in the FABQ have been correlated with changes in disability

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Virag, MPT, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Spine Physical Therapy, Madison, Wisconsin, United States

REFERENCES:
- [Result] Slater SL, Ford JJ, Richards MC, Taylor NF, Surkitt LD, Hahne AJ. The effectiveness of sub-group specific manual therapy for low back pain: a systematic review. Man Ther. 2012 Jun;17(3):201-12. doi: 10.1016/j.math.2012.01.006. Epub 2012 Mar 3. PMID 22386046
- [Result] Koumantakis GA, Watson PJ, Oldham JA. Trunk muscle stabilization training plus general exercise versus general exercise only: randomized controlled trial of patients with recurrent low back pain. Phys Ther. 2005 Mar;85(3):209-25. PMID 15733046
- [Result] Surkitt LD, Ford JJ, Hahne AJ, Pizzari T, McMeeken JM. Efficacy of directional preference management for low back pain: a systematic review. Phys Ther. 2012 May;92(5):652-65. doi: 10.2522/ptj.20100251. Epub 2012 Jan 12. PMID 22247407
- [Result] Li LC, Bombardier C. Physical therapy management of low back pain: an exploratory survey of therapist approaches. Phys Ther. 2001 Apr;81(4):1018-28. PMID 11276184
- [Result] Gore M, Tai KS, Sadosky A, Leslie D, Stacey BR. Use and costs of prescription medications and alternative treatments in patients with osteoarthritis and chronic low back pain in community-based settings. Pain Pract. 2012 Sep;12(7):550-60. doi: 10.1111/j.1533-2500.2012.00532.x. Epub 2012 Feb 5. PMID 22304678
- [Result] Rundell SD, Davenport TE. Patient education based on principles of cognitive behavioral therapy for a patient with persistent low back pain: a case report. J Orthop Sports Phys Ther. 2010 Aug;40(8):494-501. doi: 10.2519/jospt.2010.3264. PMID 20710087
- [Result] Wentz AC, Garcia SC, Klingensmith GJ, Migeon CJ, Jones GS. Gonadotropin output and response to LRH administration in congenital virilizing adrenal hyperplasia. J Clin Endocrinol Metab. 1976 Feb;42(2):239-46. doi: 10.1210/jcem-42-2-239. PMID 770494
- [Result] Flynn T, Fritz J, Whitman J, Wainner R, Magel J, Rendeiro D, Butler B, Garber M, Allison S. A clinical prediction rule for classifying patients with low back pain who demonstrate short-term improvement with spinal manipulation. Spine (Phila Pa 1976). 2002 Dec 15;27(24):2835-43. doi: 10.1097/00007632-200212150-00021. PMID 12486357
- [Result] Hicks GE, Fritz JM, Delitto A, McGill SM. Preliminary development of a clinical prediction rule for determining which patients with low back pain will respond to a stabilization exercise program. Arch Phys Med Rehabil. 2005 Sep;86(9):1753-62. doi: 10.1016/j.apmr.2005.03.033. PMID 16181938
- [Result] Fritz JM, Cleland JA, Childs JD. Subgrouping patients with low back pain: evolution of a classification approach to physical therapy. J Orthop Sports Phys Ther. 2007 Jun;37(6):290-302. doi: 10.2519/jospt.2007.2498. PMID 17612355
- [Result] Khalil H, Quinn L, van Deursen R, Dawes H, Playle R, Rosser A, Busse M. What effect does a structured home-based exercise programme have on people with Huntington's disease? A randomized, controlled pilot study. Clin Rehabil. 2013 Jul;27(7):646-58. doi: 10.1177/0269215512473762. Epub 2013 Feb 20. PMID 23426565
- [Result] Betker AL, Desai A, Nett C, Kapadia N, Szturm T. Game-based exercises for dynamic short-sitting balance rehabilitation of people with chronic spinal cord and traumatic brain injuries. Phys Ther. 2007 Oct;87(10):1389-98. doi: 10.2522/ptj.20060229. Epub 2007 Aug 21. PMID 17712036
- [Result] Murphy KM, Rasmussen L, Hervey-Jumper SL, Justice D, Nelson VS, Yang LJ. An assessment of the compliance and utility of a home exercise DVD for caregivers of children and adolescents with brachial plexus palsy: a pilot study. PM R. 2012 Mar;4(3):190-7. doi: 10.1016/j.pmrj.2011.08.538. Epub 2011 Nov 16. PMID 22088854
- [Result] Reo JA, Mercer VS. Effects of live, videotaped, or written instruction on learning an upper-extremity exercise program. Phys Ther. 2004 Jul;84(7):622-33. PMID 15225081
- [Result] Armstrong AW, Kim RH, Idriss NZ, Larsen LN, Lio PA. Online video improves clinical outcomes in adults with atopic dermatitis: a randomized controlled trial. J Am Acad Dermatol. 2011 Mar;64(3):502-7. doi: 10.1016/j.jaad.2010.01.051. Epub 2011 Jan 13. PMID 21236514
- [Result] Idriss NZ, Alikhan A, Baba K, Armstrong AW. Online, video-based patient education improves melanoma awareness: a randomized controlled trial. Telemed J E Health. 2009 Dec;15(10):992-7. doi: 10.1089/tmj.2009.0055. PMID 20028190
- [Result] O'Donnell L, San Doval A, Duran R, O'Donnell CR. The effectiveness of video-based interventions in promoting condom acquisition among STD clinic patients. Sex Transm Dis. 1995 Mar-Apr;22(2):97-103. doi: 10.1097/00007435-199503000-00004. PMID 7624818
- [Result] Hicks GE, Fritz JM, Delitto A, Mishock J. Interrater reliability of clinical examination measures for identification of lumbar segmental instability. Arch Phys Med Rehabil. 2003 Dec;84(12):1858-64. doi: 10.1016/s0003-9993(03)00365-4. PMID 14669195
- [Result] Persson AV, Frusha JD, Chevalier RJ. Rapid preparation of lecture slides. Surg Clin North Am. 1985 Feb;65(1):139-48. doi: 10.1016/s0039-6109(16)43538-3. PMID 3992439
- [Result] Inott T, Kennedy BB. Assessing learning styles: practical tips for patient education. Nurs Clin North Am. 2011 Sep;46(3):313-20, vi. doi: 10.1016/j.cnur.2011.05.006. PMID 21791266
- [Result] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Result] Jensen MP, Turner JA, Romano JM. What is the maximum number of levels needed in pain intensity measurement? Pain. 1994 Sep;58(3):387-392. doi: 10.1016/0304-3959(94)90133-3. PMID 7838588
- [Result] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Result] George SZ, Valencia C, Beneciuk JM. A psychometric investigation of fear-avoidance model measures in patients with chronic low back pain. J Orthop Sports Phys Ther. 2010 Apr;40(4):197-205. doi: 10.2519/jospt.2010.3298. PMID 20357418
- [Result] George SZ, Stryker SE. Fear-avoidance beliefs and clinical outcomes for patients seeking outpatient physical therapy for musculoskeletal pain conditions. J Orthop Sports Phys Ther. 2011 Apr;41(4):249-59. doi: 10.2519/jospt.2011.3488. Epub 2011 Feb 18. PMID 21335927
- [Result] Pfingsten M, Kroner-Herwig B, Leibing E, Kronshage U, Hildebrandt J. Validation of the German version of the Fear-Avoidance Beliefs Questionnaire (FABQ). Eur J Pain. 2000;4(3):259-66. doi: 10.1053/eujp.2000.0178. PMID 10985869
- [Result] Chaory K, Fayad F, Rannou F, Lefevre-Colau MM, Fermanian J, Revel M, Poiraudeau S. Validation of the French version of the fear avoidance belief questionnaire. Spine (Phila Pa 1976). 2004 Apr 15;29(8):908-13. doi: 10.1097/00007632-200404150-00018. PMID 15082995
- [Result] Fritz JM, George SZ. Identifying psychosocial variables in patients with acute work-related low back pain: the importance of fear-avoidance beliefs. Phys Ther. 2002 Oct;82(10):973-83. PMID 12350212
- [Result] Woby SR, Watson PJ, Roach NK, Urmston M. Adjustment to chronic low back pain--the relative influence of fear-avoidance beliefs, catastrophizing, and appraisals of control. Behav Res Ther. 2004 Jul;42(7):761-74. doi: 10.1016/S0005-7967(03)00195-5. PMID 15149897
- [Result] Fritz JM, Irrgang JJ. A comparison of a modified Oswestry Low Back Pain Disability Questionnaire and the Quebec Back Pain Disability Scale. Phys Ther. 2001 Feb;81(2):776-88. doi: 10.1093/ptj/81.2.776. PMID 11175676
- [Result] Waddell G, Somerville D, Henderson I, Newton M. Objective clinical evaluation of physical impairment in chronic low back pain. Spine (Phila Pa 1976). 1992 Jun;17(6):617-28. doi: 10.1097/00007632-199206000-00001. PMID 1308095
- [Result] Maher CG, Simmonds M, Adams R. Therapists' conceptualization and characterization of the clinical concept of spinal stiffness. Phys Ther. 1998 Mar;78(3):289-300. doi: 10.1093/ptj/78.3.289. PMID 9520974
- [Result] Nachemson AL. Advances in low-back pain. Clin Orthop Relat Res. 1985 Nov;(200):266-78. PMID 2933201
- [Result] Beurskens AJHM, de Vet HCW, Koke AJA. Responsiveness of functional status in low back pain: a comparison of different instruments. Pain. 1996 Apr;65(1):71-76. doi: 10.1016/0304-3959(95)00149-2. PMID 8826492
- See also: American Pain Foundation — http://painfoundation.org